CLINICAL TRIAL: NCT02498483
Title: Acetaminophen and Post Circumcision Pain Control
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Understaffing
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAAN7406
Record Dates: First submitted 2015-06-30; First posted 2015-07-15 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Pain; Circumcision
Keywords: Infant pain; Acetaminophen; Circumcision
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetaminophen Arm (Experimental): Acetaminophen 15 mg/kg PO solution administered via syringe one time immediately post circumcision.
  Interventions: Drug: Acetaminophen
- Non-treatment Arm (No Intervention): Routine circumcision without acetaminophen.

INTERVENTIONS:
Drug: Acetaminophen — Infants will receive 15 mg/kg of acetaminophen.
  Arms: Acetaminophen Arm

SUMMARY:
Infants do not routinely receive acetaminophen for pain control after circumcision. This study will determine if acetaminophen is effective at controlling infant pain after circumcision using nerve block and oral dextrose. Infants will undergo the routine circumcision procedure, and half will be randomly selected to receive half acetaminophen immediately at the end of the procedure. Afterwards, infant's vitals signs (heart rate, respiratory rate, oxygen saturation), the neonatal infant pain scale (NIPS), and salivary cortisol levels will be checked in regular intervals up to 4 hours. The NIPS is a validated pain scoring system based on the appearance of the infant. A reduction in NIPS for those infants who receive acetaminophen versus nothing will be the primary outcome to determine if the study is significant.

DETAILED DESCRIPTION:
Male circumcision is a common surgical procedure performed in the newborn period. The American Academy of Pediatrics Task Force on Circumcision recently published an update on circumcision policy stating the benefits of male circumcision outweigh the risks. Given this update, the investigators anticipate a percentage of families who were previously undecided about circumcision will choose to have their newborn circumcised. A common concern for both parents and physicians is effective pain control. For intra-operative pain control, dorsal penile nerve block (DPNB) has been found to be the most effective when compared to EMLA (lidocaine-prilocaine) or placebo. Acetaminophen is a relatively safe, easy to administer analgesic. Prior studies have suggested that acetaminophen could be helpful in postoperative comfort. However, studies examining the effectiveness of acetaminophen for postoperative pain control in infants who received DPNB are lacking. In addition, prior studies have been incomplete in the assessment of neonatal pain.

ELIGIBILITY:
Inclusion Criteria:

Healthy newborns between 36-42 weeks gestational age Admitted to the well baby nursery who's parents are requesting circumcision. Eligibility includes

1. Apgar score at 5 minutes >7
2. birthweight greater than 2.4 kg
3. Age of at least 10 hours
4. At least one void.

Exclusion Criteria:

1. Newborns of substance abusing mothers.
2. Newborns with any contraindications to routine circumcision, anatomical or hematologic.

Ages: 10 Hours to 36 Hours | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2015-09; Primary Completion 2017-01 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roya O'Neal, MD, Principal Investigator — Columbia University
Locations (1):
- Well Baby Nursery at New York Prebyterian-Columbia, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: Includes subjects who received acetaminophen 15 mg/kg PO solution administered via syringe one time immediately post circumcision.
- Control Arm: Includes subjects who received routine care post circumcision.
Period: Overall Study
Arm/Group | Treatment Arm | Control Arm
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control Arm | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 5 | 11
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 5 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Neonatal Infant Pain Scale (NIPS)
Description: The Neonatal Infant Pain Scale (NIPS) is a behavioral scale and can be utilized with both full-term and pre-term infants. The tool uses the behaviors that nurses have described as being indicative of infant pain or distress. It is composed of six (6) indicators: facial expression, cry, breathing patterns, arms, legs and state of arousal. Each behavioral indicator is scored with 0 or 1 except "cry", which has three possible descriptors therefore, being scored with a 0, 1 or 2. Infants are observed for one minute in order to fully assess each indicator. Total pain scores range from 0-7, with a score of 0-2 indicating mild to no pain and no suggested intervention (better outcome) to a score >4 indicating severe pain, suggesting non-pharmacological and/or pharmacological interventions may be needed.
Time Frame: Baseline and 4 hours
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Acetaminophen Arm | Non-treatment Arm
Number analyzed (Participants) | 6 | 5
score on a scale
  Baseline | 2.5 [0 to 7] | 3.2 [0 to 6]
  4 Hours post-circumcision | 1.0 [0 to 2] | 1.4 [0 to 3]

2. Secondary Outcome: Heart Rate
Time Frame: Baseline and 4 hours
Measure: Mean (Full Range); unit: Beats per minute
Arm/Group | Acetaminophen Arm | Non-treatment Arm
Number analyzed (Participants) | 6 | 5
Beats per minute
  Baseline | 138.7 [120 to 156] | 128.8 [108 to 179]
  4 Hours post-circumcision | 125 [116 to 136] | 124.8 [101 to 150]

3. Secondary Outcome: Change in Salivary Cortisol Rise
Time Frame: Baseline and 4 hours
Population: Only subjects who were able to provide saliva were incorporated into the data analysis. One subject in the acetaminophen arm could not provide a saliva sample for analysis, and 2 subjects in the control arm could not provide saliva samples for analysis.
Measure: Mean (Full Range); unit: nmol/L
Arm/Group | Acetaminophen Arm | Non-treatment Arm
Number analyzed (Participants) | 5 | 3
nmol/L
  Baseline | 0.389 [0.159 to 0.917] | 0.427 [0.171 to 0.721]
  30 minutes post-circumcision | 1.085 [0.439 to 2.779] | 0.811 [0.702 to 0.925]

4. Secondary Outcome: Respiratory Rate
Time Frame: Baseline and 4 hours
Measure: Mean (Full Range); unit: breaths per minute
Arm/Group | Acetaminophen Arm | Non-treatment Arm
Number analyzed (Participants) | 6 | 5
breaths per minute
  Baseline | 59.7 [40 to 94] | 45 [40 to 52]
  4 Hours post-circumcision | 42 [28 to 58] | 43.6 [40 to 56]

5. Secondary Outcome: Pulse Oximetry
Time Frame: Baseline 4 hours
Measure: Mean (Full Range); unit: percentage of oxygen saturation
Arm/Group | Acetaminophen Arm | Non-treatment Arm
Number analyzed (Participants) | 6 | 5
percentage of oxygen saturation
  Baseline | 98.8 [97 to 100] | 98.2 [96 to 100]
  4 Hours post-circumcision | 97.5 [96 to 100] | 98.4 [95 to 100]

ADVERSE EVENTS:
Description: The AE data is reported for the combination of all arms/groups because the data was collected and observed for the entire study population and not per arm.
Arm/Group | Acetaminophen Arm | Non-treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes